CLINICAL TRIAL: NCT00214370
Title: Propofol Versus Propofol-Fentanyl as Sedation For Lumbar Puncture in Children With Acute Leukemia/Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-0470
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2007-07

CONDITIONS: Leukemia; Lymphoma
Keywords: pediatric; acute leukemia/lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Propofol

INTERVENTIONS:
Drug: Propofol-Fentanyl
Drug: Propofol alone

SUMMARY:
The hypothesis of the study is that propofol-fentanyl sedation for lumbar punctures in children with acute leukemia/lymphoma results in fewer adverse events than propofol sedation alone. Secondary hypotheses state that propofol-fentanyl sedation results in a better sedation induction, recovery profile and is preferred by patients/families. The study is a double blind, randomized, placebo controlled crossover study. Following the induction phase of chemotherapy, children will be randomized in a crossover manner to receive either fentanyl-propofol or propofol-placebo for future lumbar punctures. Patients will be studied on two separate occasions, once with propofol-placebo (normal saline) and once with propofol-fentanyl. Children will be monitored continuously by pulse oximetry, electrocardiogram (ECG) and direct nursing and physician observation during the sedation in accordance with the University of Wisconsin (UW) Pediatric Policy and Procedure. Propofol will be titrated to a Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) score of ≤ 7 for all children. Oxygen saturation, respiratory rate, heart rate and blood pressure will be recorded every 3 minutes by a study investigator during sedation.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2 years to 18 years with acute leukemia/lymphoma cared for by physicians in the Division of Hematology/Oncology in the Department of Pediatrics and receiving sedation for diagnostic/therapeutic lumbar punctures (LPs) in the UW Pediatric Sedation Program
* Enrollment will occur after the induction phase of chemotherapy.

Exclusion Criteria:

* American Society of Anesthesiology score ≥ 3
* Cardiorespiratory instability
* Allergy to propofol or its components
* Age less than 2 years
* Patients receiving other sedative analgesics
* Patients with an oxygen requirement

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Fewer adverse cardiorespiratory events defined as oxygen desaturations and hypotension

SECONDARY OUTCOMES:
Patient/family preference, ease of induction, and recovery pattern

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hollman, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States